CLINICAL TRIAL: NCT05912660
Title: Health Status of Patients After Surgically Implanted Biological and TAVI: a Population-based Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Sicknessfund Burgenland (Unknown); Landesklinikum Sankt Polten (Other)
Responsible Party: Principal Investigator, Hendrik Jan Ankersmit, Univ. Prof. , MD, MBA, Medical University of Vienna
Other Study IDs: AUTHEARTVISIT - TAVI
Record Dates: First submitted 2023-06-10; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Aortic valve replacement with surgically implanted bioprostheses
  Interventions: Device: Aortic Valve Replacement
- Aortic valve replacement with TAVI
  Interventions: Device: Aortic Valve Replacement

INTERVENTIONS:
Device: Aortic Valve Replacement — Aortic Valve Replacement (surgically or TAVI)

SUMMARY:
The overall project aim is to study outcomes following aortic valve replacement with surgically implanted bioprostheses or TAVI by retrieving data from the main social security carriers in Austria for the years 2010-2020.

ELIGIBILITY:
Inclusion Criteria:

* isolated aortic valve replacement in Austria (surgically implanted bioprostheses or TAVI)

Exclusion Criteria:

* below 65 years of age
* coronary revascularization within 4 months before the index procedure
* concomitant heart surgery

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients who underwent isolated aortic valve replacement in Austria (surgically implanted bioprostheses or TAVI) above 65 years of age with no other concomitant heart surgery and no coronary revascularization within 4 months before the index procedure were included.
Sampling Method: Non-Probability Sample
Enrollment: 18882 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 10 years
  all cause mortality after aortic valve replacement

SECONDARY OUTCOMES:
reoperation | 10 years
  incidence of reoperation after aortic valve replacement
myocardial infaction | 10 years
  incidence of myocardial infaction after aortic valve replacement
heart failure | 10 years
  incidence of heart failure after aortic valve replacement
stroke | 10 years
  incidence of stroke after aortic valve replacement

IPD SHARING:
Plan to Share IPD: No